CLINICAL TRIAL: NCT05924269
Title: Role of Neuronal Guidance Proteins as Diagnostic Markers for Acute Kidney Injury (AKI)
Acronym: NEUKID
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: NEUKID
Record Dates: First submitted 2023-06-20; First posted 2023-06-29 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Acute Kidney Injury
Keywords: Neuronal Guidance Protein; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Surgery: Patients undergoing cardiac surgery

SUMMARY:
Acute kidney failure remains one of the most challenging entities to diagnose in clinical medicine, especially in the field of intensive care. The diagnosis of acute kidney injury is based solely on urine output and serum creatinine, both of which could also be influenced by other factors. A more sensitive and faster diagnostic option would not only be desirable but of utmost clinical importance. Therefore, the investigators aim to identify Neuronal Guidance Proteins (NGPs) as potential biomarkers for the identification and early detection of AKI with this investigation. This investigation aims to identify the possibility of diagnosing acute kidney injury, the subsequent validation of a potential biomarker will then have to take place in a multicenter study approach: Data in preclinical mouse models suggest that SEMA7A as one of the NGPs could be valuable as a biomarker, the study now aims to attempt a preliminary survey in humans and measure various NGPs.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery
* written consent

Exclusion Criteria:

* no written consent possible
* Polytrauma, severe burns
* Immunosuppression
* Pregnancy
* Diagnosis of Hepatitis B, Hepatitis C, and/or HIV
* Sepsis
* Pre-existing kidney damage

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective cardiac surgery followed by postoperative surveillance in the intensive care unit
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
AKI | 1-7 days
  Development of AKI after cardiac surgery

SECONDARY OUTCOMES:
NGP | 1-7 days
  Concentration of NGPs in Blood and Urine

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Körner, MD, Principal Investigator — University Clinic of Tuebingen

IPD SHARING:
Plan to Share IPD: No